CLINICAL TRIAL: NCT04165486
Title: A Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of ION464 Administered Intrathecally to Adults With Multiple System Atrophy
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ION464 Administered to Adults With Multiple System Atrophy (HORIZON)
Acronym: HORIZON
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ION464-CS1; 2019-001105-24 (EudraCT Number)
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: ION464 (Experimental): ION464 will be administered at multiple-ascending doses by IT injection at regular intervals over 12 weeks.
  Interventions: Drug: ION464
- Part 1: Placebo (Placebo Comparator): ION464-matching placebo will be administered by IT injection at regular intervals over 12 weeks.
  Interventions: Drug: Placebo
- Part 2: ION464 (Experimental): ION464 will be administered at the same doses as Part 1 by IT injection, at regular intervals, for 72 weeks.
  Interventions: Drug: ION464
- Part 2: Placebo (Placebo Comparator): ION464-matching placebo will be administered by IT injection, at regular intervals, for 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ION464 — ION464 will be administered by IT injection.
  Arms: Part 1: ION464; Part 2: ION464
Drug: Placebo — ION464-matching placebo will be administered by IT injection.
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
The primary objectives are to evaluate the safety and tolerability of multiple doses of ION464 administered via intrathecal (IT) injection (Part 1) and to evaluate the long-term safety and tolerability of ION464 (Part 2) in participants with multiple system atrophy (MSA).

The secondary objectives are to evaluate the pharmacodynamic (PD) effect of ION464 on the level of a potential biomarker of target engagement (Parts 1 and 2) and to evaluate the pharmacokinetic (PK) profile of ION464 in serum (Part 1).

DETAILED DESCRIPTION:
This is a first-in-human, randomized, blinded, placebo-controlled, multiple-ascending-dose (MAD) study (Part 1) to evaluate the safety, tolerability, PK, and PD of ION464 in adult participants diagnosed with MSA with a long-term extension (LTE) (Part 2). The study will include up to approximately 40 participants. Part 1 of the study consists of a Screening Period of up to 6 weeks, a Treatment Period of 12 weeks, and a Follow-up Period of 24 weeks. The study duration for each participant in Part 2 will be approximately 96 weeks, which consists of a 72-week Treatment Period and a 24-week Follow-up Period.

ELIGIBILITY:
Key Inclusion Criteria:

* Screening single-photon emission computed tomography (SPECT) with DaTscan™ (ioflupane I123 injection) results demonstrating loss (whether symmetric or asymmetric) of dopamine nerve terminals in the striatum consistent with neurodegenerative parkinsonism, as assessed with qualitative, visual read.
* Diagnosed with probable or possible MSA, either parkinsonian-type (MSA-P) or cerebellar-type (MSA-C).
* Must be able to walk unassisted for at least 10 meters (approximately 30 feet)

Key Exclusion Criteria:

* Presence of cognitive dysfunction (defined as Montreal Cognitive Assessment (MoCA) score <25)
* Family history of ataxia or parkinsonism and known genetic cause of ataxia or parkinsonism.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Baseline up to approximately 36 weeks
Number of Participants with Serious Adverse Events (SAEs) | Baseline up to approximately 36 weeks

SECONDARY OUTCOMES:
Change From Baseline in Cerebrospinal Fluid (CSF) Levels of Total alpha-synuclein (α-syn) | Baseline up to approximately 36 weeks
Serum Concentration of ION464 | Baseline up to approximately 36 weeks
Area Under the Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration of ION464 | Baseline up to approximately 36 weeks
Maximum Observed Concentration (Cmax) of ION464 | Baseline up to approximately 36 weeks
Time to Reach Maximum Observed Concentration (Tmax) of ION464 | Baseline up to approximately 36 weeks

CONTACTS AND LOCATIONS:
Locations (14):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- France (3):
  - CHU de Lyon - Hospices Civils de Lyon-H6pital Pierre Wertheimer, Neurologique HCL, Lyon
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hopital Purpan, Toulouse
- Germany (5):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf
  - Medizinische Hochschule Hannover (MHH), Hanover
  - University Hospital Marburg, Marburg
  - Klinikum der Universtiatet Muenchen -Campus Grosshadern, München
- Hospital Beatriz Ângelo, Loures, Portugal
- United Kingdom (4):
  - Institute of Neurology & The National Hospital for Neurology and Neurosurgery, London, England
  - The John Radcliffe Hospital, Oxford, England
  - Salford Royal Hospital, Salford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No